CLINICAL TRIAL: NCT05770856
Title: Clinical Metagenomic Next-Generation Sequencing for Microbial Infections in Trauma
Brief Title: Clinical Metagenomic of Post-traumatic Infections
Acronym: METADIAG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Military Teaching Hospital Sainte Anne, Toulon (Unknown); UMR Vitrome, IRD 257 (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-CHITS-003
Record Dates: First submitted 2023-02-07; First posted 2023-03-16 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Fractures, Bone; Infections
Keywords: High throughput sequencing; Nanopore; Diagnosis; Trauma; Microbiome; Infection
MeSH Terms: conditions — Fractures, Bone; Infections; Disease; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Surgical bone and soft tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma related infection
  Interventions: Diagnostic Test: Metagenomic sequencing

INTERVENTIONS:
Diagnostic Test: Metagenomic sequencing — Samples shall be submitted to high throughput sequencing using both illumine MiSeq and Oxford Nanopore Technologies.

SUMMARY:
Treatment of fracture related infection is challenging and often lead to failure in such situation that carry a high health cost burden.

These infections are often polymicrobial, making the identification of all involved microorganisms a major concern to provide tailored antibiotic treatment. Culture-independent methods are needed to better represent the microbial diversity of infected wounds. Metagenomic sequencing might lead to an accurate microbiome characterization in infected trauma-related wound.

Preliminary studies have reported results of metagenomic sequencing in diabetic foot infection but data focusing on non-diabetic infected patients are scarce.

The impact of post-traumatic infected wound microbiome needs to be assessed, with regards to bacterial abundance, diversity including at the strain level and functional genes, along with their longitudinal evolution and association with clinical outcomes.

DETAILED DESCRIPTION:
DNA will be extracted from samples carried out during surgical procedures. Different extraction protocols will be assessed to determine the best to be used for this type of tissue samples.

Purified DNA will be quantified using the Qubit dsDNA High-Sensitivity Assay Kit (Invitrogen). The quality of the fragment length will be estimated with the DNA high-sensitivity kit in the 2100 Bioanalyzer (Agilent Technologies). DNA sequencing will be performed with Oxford Nanopore Technologie devices: MinIONTM and GridIONTM.

Another sequencing of the same samples will be performed on the MiSeq after libraries preparation using the NexteraXT DNA Library Preparation Kit (Illumina).

Sequenced OTU from both sequencing methods will be confronted at different taxonomic ranks and compared with conventional routine method results (bacterial culture). A functional analysis of sequences will be done to identify potential genes associated with clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of trauma-related infection

Exclusion Criteria:

* Participation in an interventional research during the study
* Patient opposition
* Absence of bone or soft tissue samples stored at -80°C

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital for trauma for which an infection of the traumatic site was diagnosed
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Microbiome of fracture-related and other trauma-related infection | About 2 months
  Metagenomic sequencing will be used to determine the microbiome of trauma-related infections using Illumina MiSeq and Oxford Nanopore Technologies.
  Data will be compared with those from reference microbiological identification techniques (culture).

SECONDARY OUTCOMES:
Comparison of high throughput sequencing techniques yield | About 3 months
  The FRI-associated microbiomes composition obtained with each sequencing methods will be compared in terms of abundance and variety (K coefficient and frequency)
Number and nature of virulence or resistance factors among identified OTU (operational Taxonomic Unit) | About 6 months
  Functional annotation of sequenced bacterial genomes to assess the presence of virulence and/or resistance-associated factors, using Prokka software.
Number of bacteria and their relative abundance according to patients' outcome using the EBJIS (European Bone and Joint Infection) definition | About 6 months
  To determine the association of the NGS-based microbiome longtitudinal composition in terms of variety (number of OTU) and abundance (number of reads) with infection persistence according to the EBJIS (European Bone and Joint Infection) definition.

CONTACTS AND LOCATIONS:
Overall Officials: David LACÔTE-DELARBRE, MD, Study Director — Military Teaching Hospital Sainte Anne
Locations (1):
- Military Teaching Hospital Sainte Anne, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ivy MI, Thoendel MJ, Jeraldo PR, Greenwood-Quaintance KE, Hanssen AD, Abdel MP, Chia N, Yao JZ, Tande AJ, Mandrekar JN, Patel R. Direct Detection and Identification of Prosthetic Joint Infection Pathogens in Synovial Fluid by Metagenomic Shotgun Sequencing. J Clin Microbiol. 2018 Aug 27;56(9):e00402-18. doi: 10.1128/JCM.00402-18. Print 2018 Sep. PMID 29848568
- [Background] Jnana A, Muthuraman V, Varghese VK, Chakrabarty S, Murali TS, Ramachandra L, Shenoy KR, Rodrigues GS, Prasad SS, Dendukuri D, Morschhauser A, Nestler J, Peter H, Bier FF, Satyamoorthy K. Microbial Community Distribution and Core Microbiome in Successive Wound Grades of Individuals with Diabetic Foot Ulcers. Appl Environ Microbiol. 2020 Mar 2;86(6):e02608-19. doi: 10.1128/AEM.02608-19. Print 2020 Mar 2. PMID 31924616
- [Background] Kalan LR, Meisel JS, Loesche MA, Horwinski J, Soaita I, Chen X, Uberoi A, Gardner SE, Grice EA. Strain- and Species-Level Variation in the Microbiome of Diabetic Wounds Is Associated with Clinical Outcomes and Therapeutic Efficacy. Cell Host Microbe. 2019 May 8;25(5):641-655.e5. doi: 10.1016/j.chom.2019.03.006. Epub 2019 Apr 18. PMID 31006638
- [Background] Mudrik-Zohar H, Carasso S, Gefen T, Zalmanovich A, Katzir M, Cohen Y, Paitan Y, Geva-Zatorsky N, Chowers M. Microbiome Characterization of Infected Diabetic Foot Ulcers in Association With Clinical Outcomes: Traditional Cultures Versus Molecular Sequencing Methods. Front Cell Infect Microbiol. 2022 Mar 24;12:836699. doi: 10.3389/fcimb.2022.836699. eCollection 2022. PMID 35402307
- [Result] Delarbre D, Lavrard P, Elias A, Bossi V, Kacel I, Janvier F, Fournier PE. Bacterial DNA enrichment for low-inoculum fracture-related infection diagnostic using high-throughput sequencing. Diagn Microbiol Infect Dis. 2024 Sep;110(1):116411. doi: 10.1016/j.diagmicrobio.2024.116411. Epub 2024 Jun 22. PMID 39018934